CLINICAL TRIAL: NCT06793527
Title: Comparison of the Efficacy of Celiac Plexus Blockade, Erector Spinae Compartment Blockade (ESP), and Intravenous Lidocaine Infusion Under Opioid-free Anesthesia in Patients Undergoing Bariatric Surgery
Brief Title: Comparison of the Efficacy of Celiac Plexus Blockade, ESP and Lidocaine Infusion Under OFA
Acronym: LECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, MD PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1072.6120.116.2024
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Regional Anaesthesia; Anesthesia and Analgesia
Keywords: ESP; celiac plexus block; OFA; erector spinal plane block; opioid free anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinal BLock (Experimental): Before the procedure, a block of the erector spinae (ESP) compartment will be performed with approximately 20 ml of 0.25% ropivacaine at the Th4 level. The patient will be informed about the possibility of short-term discomfort if the block is performed before full induction of anesthesia.
  Interventions: Drug: ESP block
- Celiac Plexus Block (Experimental): During general anesthesia, a celiac plexus block will be performed intraoperatively (20 ml of 0.5% ropivacaine). The patient will not feel discomfort due to general anesthesia.
  Interventions: Drug: Celiac Plexus Block
- Lidocaine IV (Placebo Comparator): Instead of a regional block, an intravenous infusion of lidocaine will be used.
  Interventions: Drug: Lidacaine

INTERVENTIONS:
Drug: Celiac Plexus Block — During general anesthesia, a celiac plexus block will be performed intraoperatively (20 ml of 0.5% ropivacaine). The patient will not feel discomfort due to general anesthesia.
  Arms: Celiac Plexus Block
Drug: ESP block — Before the procedure, a block of the erector spinae (ESP) compartment will be performed with approximately 20 ml of 0.25% ropivacaine at the Th4 level. The patient will be informed about the possibility of short-term discomfort if the block is performed before full induction of anesthesia.
  Arms: Erector Spinal BLock
Drug: Lidacaine — Instead of a regional block, an intravenous infusion of lidocaine will be used.
  Arms: Lidocaine IV

SUMMARY:
Modern anesthesiology, in search of alternatives to opioid-based pain management, is turning to low-opioid and non-opioid protocols. Replacing opioids with non-opioid analgesics, co-analgesics, and regional and local anesthesia techniques allows avoiding the adverse effects of opioids while maintaining satisfactory analgesia. This is of particular importance in bariatric surgery, where reducing the incidence of respiratory depression, sedation, opioid hyperalgesia, and postoperative nausea and vomiting is a priority. Standard non-opioid anesthesia (OFA) includes ketamine, lidocaine, and dexmedetomidine infusions, while regional techniques additionally reduce the need for analgesics. Despite the widespread use of these methods, there is no clear data on the superiority of any of them in bariatric procedures.

DETAILED DESCRIPTION:
This is a prospective, randomized study with random assignment of patients to three groups:

ESP group: Before the procedure, a block of the erector spinae (ESP) compartment will be performed with approximately 20 ml of 0.25% ropivacaine at the Th4 level. The patient will be informed about the possibility of short-term discomfort if the block is performed before full induction of anesthesia.

Celiac plexus group: During general anesthesia, a celiac plexus block will be performed intraoperatively (20 ml of 0.5% ropivacaine). The patient will not feel discomfort due to general anesthesia.

Lidocaine IV group: Instead of a regional block, an intravenous infusion of lidocaine will be used.

All three methods are recognized methods of perioperative anesthesia. There is no placebo group in the study - intravenous infusion of lidocaine is the reference method, and both regional blocks are compared in relation to it and to each other.

All groups will be anesthetized without opioids using ketamine, dexmedetomidine and inhaled sevoflurane. After surgery, patients will receive standard analgesic therapy (oxycodone with naloxone, paracetamol, metamizole, dexketoprofen). They will be informed about the possible side effects of opioids, although the main goal is to minimize their use during the procedure.

Pain intensity will be assessed using the NRS scale at 1, 2, 6, 12 and 24 hours after the procedure. In addition, on the postoperative day, the patient will complete the QOR-15 questionnaire, and the frequency of postoperative nausea and vomiting will also be monitored.

The choice of ropivacaine is due to its more favorable cardiotoxicity profile compared to bupivacaine. The exclusion criteria will include, among others, patients taking medications that may increase the risk of arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years who underwent laparoscopic bariatric surgery
* Must be able to sign agreement for study

Exclusion Criteria:

* Patients with a history of allergic reactions to drugs
* Patients with a history of drug addiction
* Patients with chronic pain who require analgesics
* History of hospitalization for psychiatric disorders
* Preoperative pulse oximetry (SpO2) < 95 %
* bradycardia (HR<50bpm)
* hypotension
* atrioventricular block
* intraventricular or sinus block
* Blood clotting disorders
* Pregnant/lactating women
* Cognitive impairment
* Unable to read consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Life quality | 1 day
  Every patient will do OR-15

SECONDARY OUTCOMES:
posoperative pain | 1 day
  NRS score after operation from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skladzien, MD PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Department of Intensive Interdisciplinary Care, Collegium Medicum, Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Our patients do not agree on share their data

REFERENCES:
- [Result] Hung KC, Chiu CC, Hsu CW, Lin CM, Liao SW, Teng IC, Chen IW, Sun CK. Impact of Opioid-Free Anesthesia on Analgesia and Recovery Following Bariatric Surgery: a Meta-Analysis of Randomized Controlled Studies. Obes Surg. 2022 Sep;32(9):3113-3124. doi: 10.1007/s11695-022-06213-7. Epub 2022 Jul 19. PMID 35854095